CLINICAL TRIAL: NCT00737945
Title: Incremental Significance of Endothelial Function Assessed by Reactive Hyperemia Peripheral Arterial Tonometry to Improve Risk Stratification in High Risk Patients for Cardiovascular Events
Brief Title: Prognostic Value of Endothelial Dysfunction and Coronary Complexity
Status: Completed | Type: Observational
Sponsor: Kumamoto University (Other)
Responsible Party: Principal Investigator, Seigo Sugiyama, Department of Cardiovascular Medicine, Kumamoto University
Other Study IDs: 0804
Record Dates: First submitted 2008-08-18; First posted 2008-08-20 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 2

SUMMARY:
The investigators test the additional clinical value of the physiological assessment of endothelial function to the morphological assessment of coronary complexity and classical risk score in predicting cardiovascular events.

DETAILED DESCRIPTION:
The investigators enroll consecutive, stable high risk patients for cardiovascular events. The reactive hyperemia peripheral arterial tonometry index (RHI) was measured before coronary angiography and coronary lesions were assessed angiographically by SYNTAX Scoring system. The investigators all subjects and examined the occurrence of cardiovascular events (CV death, non-fatal myocardial infarction and ischemic stroke, unstable angina pectoris, hospitalization for HF, coronary revascularization, or non-fatal aortic and peripheral vascular disease).

ELIGIBILITY:
Inclusion Criteria:

* Stable, high-risk patients with diabetes mellitus, or more than two conventional coronary risk factors, who are referred for coronary angiography because of angina-like chest symptoms.

Exclusion Criteria:

* An ejection fraction < 50%
* Moderate to severe valvular heart disease
* Cardiomyopathy
* Allergy to latex
* Significant endocrine, hepatic, renal, or inflammatory disease
* cerebrovascular disease

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kumamoto University Hospital and Yokohama City University Medical Center
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2006-08; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Cardiovascular event | Outcome is assessed 1 to 4 years after entry
  Cardiovascular event consists of cardiovascular death, myocardial infarction, unstable angina, ischemic stroke, coronary revascularization, hospitalization for heart failure, aortic disease and peripheral arterial disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Kumamoto University Hospital, Kumamoto, Japan

REFERENCES:
- [Derived] Matsuzawa Y, Sugiyama S, Sumida H, Sugamura K, Nozaki T, Ohba K, Matsubara J, Kurokawa H, Fujisue K, Konishi M, Akiyama E, Suzuki H, Nagayoshi Y, Yamamuro M, Sakamoto K, Iwashita S, Jinnouchi H, Taguri M, Morita S, Matsui K, Kimura K, Umemura S, Ogawa H. Peripheral endothelial function and cardiovascular events in high-risk patients. J Am Heart Assoc. 2013 Nov 25;2(6):e000426. doi: 10.1161/JAHA.113.000426. PMID 24275629